CLINICAL TRIAL: NCT04652518
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Trial and Open Label Extension to Evaluate the Safety and Efficacy of Deupirfenidone (LYT-100) in Post-acute COVID-19 Respiratory Disease
Brief Title: LYT-100 in Post-acute COVID-19 Respiratory Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Part A of the study was completed; Part B of the study was terminated
Sponsor: PureTech (Industry)
Collaborators: Clinipace Worldwide (Industry); Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LYT-100-2020-02
Record Dates: First submitted 2020-12-02; First posted 2020-12-03 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-10

CONDITIONS: Covid19; Post-acute COVID-19 Respiratory Disease
Keywords: COVID-19 Respiratory Disease; novel coronavirus; respiratory complications; SARS-CoV-2; post acute; lung fibrosis; interstitial lung disease; long COVID; long haul COVID; Post-acute COVID-19 Respiratory Disease
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis; Lung Diseases, Interstitial; Post-Acute COVID-19 Syndrome | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LYT-100 (Experimental): LYT-100 taken orally twice a day (BID) for 91 days
  Interventions: Drug: LYT-100
- Placebo (Placebo Comparator): Placebo matching LYT-100 taken orally BID for 91 days
  Interventions: Other: Placebo
- Open Label Extension LYT-100 (Other): Open Label Extension: LYT-100 taken orally BID for 91 days The Open Label Extension (Part B) was terminated after results of the Double Blind Portion.
  Interventions: Drug: LYT-100

INTERVENTIONS:
Drug: LYT-100 — oral administration
  Other Names: Deupirfenidone
  Arms: LYT-100; Open Label Extension LYT-100
Other: Placebo — oral administration
  Arms: Placebo

SUMMARY:
This study is being conducted in two parts, A and B. Part A is a randomized, double-blind, parallel arm study to evaluate the safety and efficacy of LYT-100 compared to placebo in adults with post-acute COVID-19 respiratory complications. Part B is an Open Label Extension (OLE) study for patients who complete Part A.

DETAILED DESCRIPTION:
Part A of this study is a randomized, double-blind, parallel arm study being conducted at approximately 35 centers globally to evaluate the safety and efficacy of LYT-100 compared to placebo in 168 adults with post-acute COVID-19 respiratory complications who were treated with mechanical ventilation, extracorporeal membrane oxygenation, non-invasive ventilation (eg CPAP or BiPAP), high-flow nasal oxygen therapy or any other means of oxygen administration in the hospital for at least 1 day and have required only low flow nasal oxygen or no oxygen supplementation for at least 72 hours prior to screening. LYT-100 or placebo will be taken daily for up to 91 days with the primary outcome of change in distance walked on the six-minute walk test performed in line with the American Thoracic Society Respiratory Society Guidelines assessed at Day 91. Secondary endpoints, including pharmacokinetics, inflammatory biomarkers, imaging, and patient-reported outcomes of dyspnea and the 36-Item Short Form Health Survey will also be evaluated.

The second part of the study, Part B, is an open-label extension in which eligible patients who completed Part A will be enrolled and treated with open-label LYT-100 for an additional 91 days. The primary endpoint for Part B of the study is to assess the longer-term safety, tolerability, and efficacy of LYT-100 through up to 182 days of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Positive result of a molecular RT-qPCR diagnostic test or SARS-CoV-2 RNA result from a clinical specimen deemed clinically associated with the current episode of illness, warranting hospital admission as per investigator's judgement, or previously hospitalized (central and/or local laboratory COVID-19 test results are accepted from any biological material source)
* Hospitalization for COVID-19 respiratory disease and treated with supplemental oxygen (including MV, ECMO or any other means of oxygen administration) in hospital for at least 1 day
* COVID-19 pneumonia findings on imaging (chest X-ray or CT Scan) with a minimum of two lung lobes involvement
* Able to bear weight and ambulate a minimum of 10 m distance (use of inhaled oxygen permitted)
* Shortness of breath ≥ grade 3 on mBDS dyspnea scale and not requiring MV, ECMO, NIV, and/or HFNO (nasal O2 is allowed) for at least 72 hours before screening

Key Exclusion Criteria:

* Pre-existing chronic respiratory condition(s), obstructive or restrictive, for which the patient is actively taking concomitant medication are excluded. Patients with history of Idiopathic Pulmonary Fibrosis (IPF), lung cancer, pulmonary arterial hypertension, other interstitial lung diseases, severe cardiac insufficiency (grade IV) are excluded irrespective of whether they are actively being medicated for those conditions or not.
* Pre-existing co-morbid conditions preventing outcome assessments, e.g., neurological, medical, orthopedic injury/disability, disease or condition that would prevent ability to transfer and walk for 6 minutes, prior to confirmed COVID-19 diagnosis
* Unstable angina or myocardial infarction in the last month prior to screening
* Patients on MV, ECMO, NIV, and/or HFNO within the last 72 hours prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Change in distance walked on the six-minute walk test (6MWT) | Baseline to Day 91
  The 6MWT is a validated endpoint commonly used in clinical trial research

SECONDARY OUTCOMES:
Change in Dyspnoea-12 score | Baseline to Day 91
  Dyspnoea-12 measures "breathlessness severity" without reference to current activity and was developed for use in interstitial lung disease and COPD current experience ("these days.") The tool generates a total score using 12 descriptor items including seven physical and five affective items with response options none (0), mild (1), moderate (2) or severe (3). The total score ranges from 1 to 36 whereby the higher score correlates with greater breathlessness severity.
Change in Saint George Respiratory Questionnaire-I (SGRQ-I) score | Baseline to Day 91
  Saint George Respiratory Questionnaire-I (SGRQ-I) is an idiopathic pulmonary fibrosis disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with interstitial lung disease. There are 34 self-completed items with 3 domain component scores (Symptoms, Activities, and Impacts), with higher scores indicating more limitations.
Change in Modified Borg Dyspnoea Scale (mBDS) score | Baseline to Day 91
  The mBDS is an assessment tool that analyzes breathlessness under exertion. It starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal.
Quality of Life assessment as collected using the SF-36 | Baseline to Day 91
  The SF-36 (v2) is a self-administered questionnaire containing 36 items that measures functional status, well-being and overall evaluation of health in 8 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Toby Maher, MD, Principal Investigator — Keck School of Medicine, University of Southern California
Locations (31):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - North Alabama Medical Center, Florence, Alabama
  - University of Southern California - Keck School of Medicine, Los Angeles, California
  - Vista Health Research, Miami, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Coastal Pulmonary and Critical Care, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Center for Advanced Research and Education, Gainesville, Georgia
  - GenHarp Clinical Solutions, Evergreen Park, Illinois
  - Circuit Clinical/Crystal Run Healthcare LLP, Middletown, New York
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Affinity Health Corp, Nashville, Tennessee
  - Frostwood Family Medicine, Houston, Texas
  - The University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
- Argentina (3):
  - Clinica Central S.A, Villa Regina, Río Negro Province
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán, Tucumán Province
- Brazil (3):
  - CETI - Centro de Estudos em Terapias Inovadoras, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto de Doencas do Torax, Rio de Janeiro
- PMSI Republican Clinical Hospital "T. Mosneaga", Chisinau, Moldova
- Philippines (2):
  - University of the Philippines Manila - Philippine General Hospital (PGH), Manila
  - Quirino Memorial Medical Center (QMMC), Quezon City
- Romania (4):
  - National Institute for Infectious Diseases "Prof. Dr. Matei Balş" (Arensia Eploratory Medicine), Bucharest
  - Spitalul Clinic De Pneumoftiziologie "Leon Daniello" Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Dr. Victor Babes Craiova, Craiova
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Dr. Victor Babes - Timisoara, Timișoara
- Medical Center of Limited Liability Company "Harmoniya krasy", Kiev, Ukraine
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust - St Thomas' Hospital, London
  - St George's University Hospitals NHS Foundation Trust - St George's Hospital, London

REFERENCES:
- [Derived] Kulkarni T, Santiaguel J, Aul R, Harnett M, Krop J, Chen MC, Graham CS, Maher TM. Deupirfenidone (LYT-100) in post-acute sequelae of SARS-CoV-2 with respiratory complications. ERJ Open Res. 2025 Jul 21;11(4):01142-2024. doi: 10.1183/23120541.01142-2024. eCollection 2025 Jul. PMID 40692836